CLINICAL TRIAL: NCT00378950
Title: Health Literacy and Self-Management in Heart Failure
Brief Title: Educational Program for Various Health Literacy Levels to Improve the Health of Individuals With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 439; R01HL081257-01A1 (NIH)
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2016-05

CONDITIONS: Heart Failure, Congestive
Keywords: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will receive a 1-hour education session about CHF, symptom recognition, diet, exercise, and daily check ups.
  Interventions: Behavioral: Brief Educational Intervention (BEI)
- 2 (Experimental): Participants will receive a 1-hour education session about CHF, symptom recognition, diet, exercise, and daily check ups, as well as additional information on diuretic self adjustment. This group will then get several follow-up phone calls over the course of the year to reinforce these topics and help them master the knowledge and encourage behavior and lifestyle changes to align with these topics.
  Interventions: Behavioral: Teach to Goal (TTG)

INTERVENTIONS:
Behavioral: Teach to Goal (TTG) — The TTG program includes the Brief Educational Intervention (BEI) educational intervention, as well as education about diuretic self adjustment. In addition, follow-up phone calls are given to the TTG group to further reinforce the initial training and provide further training so participants will master the task.
  Other Names: TTG
  Arms: 2
Behavioral: Brief Educational Intervention (BEI) — The BEI is a one hour educational session on CHF, symptom recognition, diet, exercise, and daily checkups.
  Other Names: BEI
  Arms: 1

SUMMARY:
Heart failure (HF) affects 5 million people in the United States. Health literacy, which is the ability to read and comprehend important medical information, plays an important role in the health of individuals with HF. This study will evaluate the effectiveness of an educational program developed for various levels of health literacy at improving medical outcomes and quality of life in individuals with HF.

DETAILED DESCRIPTION:
HF is a complicated disease that often requires individuals to carefully monitor their condition. Individuals with HF must follow strict medication regimens, adhere to diet and exercise recommendations, and closely monitor symptoms and changes in weight. Individuals with low health literacy skills may have a harder time comprehending medication dosing instructions, educational materials, and the overall complexity of managing HF than individuals with higher health literacy skills. Programs that focus on building self-care skills have been proven to reduce the rate of hospitalizations among individuals with HF; only one study, however, has specifically examined the importance of health literacy in the effectiveness of these programs. Teach to Goal (TTG), a program that focuses on developing self-care skills while incorporating medical information for various health literacy levels, may improve medical outcomes in individuals with HF. The purpose of this study is to evaluate the effectiveness of TTG at improving hospitalization and death rates, quality of life, and self-care behaviors among individuals with HF.

This 1-year study will enroll individuals with HF. Eligible participants will attend a baseline study visit and complete survey questionnaires. Participants will then be randomly assigned to either TTG or a control group. The TTG group will partake in a 30- to 60-minute educational session, which will focus on improving self-care skills. They will also receive literacy-sensitive printed materials about monitoring body weight and swelling in the legs, medication administration, and a sodium reduction and exercise plan. Control group participants will partake in a shorter educational session and will receive fewer printed materials. All participants will be provided with a digital scale to self-monitor their weight at home. The TTG group will receive follow-up phone calls on Days 3, 7, 14, 21, and 28, during which study staff will assess participants' progress and will provide additional support and training as necessary. Both groups will receive phone calls at Months 1, 6, and 12. During these calls, number of hospitalizations, quality of life, and changes in self-care behavior and knowledge will be evaluated, but participants will not receive any additional training.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HF
* Currently prescribed a Loop diuretic medication
* At least one of the following findings:

  1. Chest x-ray consistent with HF (current or past x-ray with probable or definite pulmonary edema)
  2. Reduced ejection fraction on echocardiogram (ECHO), multiple gate acquisition scan (MUGA), or cardiac catheterization (less than 50%)
  3. Left ventricular hypertrophy (LVH) or diastolic filling pattern on ECHO
  4. Elevated B-type natriuretic peptide
* Currently experiencing New York Heart Association Class II-IV symptoms or has experienced these symptoms in the 6 months prior to study entry
* Has a working telephone
* Speaks English or Spanish

Exclusion Criteria:

* Patients will be ineligible if they meet ONE the following criteria:

  1. Sight - Inability to see printed educational material well enough to utilize it
  2. Cognition - Moderate to severe dementia (If medical notes state "Severe Dementia" or as determined by administering the study's cognitive screener)
  3. Surgery -Valuvular disease rated as severe (mitral stenosis, aortic stenosis or aortic regurgitation) or valuvular surgery planned within a year (i.e., bypass, angioplasty, valve replacement, heart transplant)
  4. Terminal Illness - Possessing a terminal illness with prognosis of 1 year or less
  5. Dialysis - Currently on dialysis or anticipated to start dialysis within 1 year
  6. Oxygen Dependant - Using concentrate oxygen intermittent or continuously for COPD
  7. Management of Care - Not able to control medications
  8. Other Studies -Patient enrolled (past or present) in another study where intervention status would interfere with pure outcome of this or other study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2007-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
All cause hospitalization | Measured at 12 months
All cause mortality | Measured at 12 months

SECONDARY OUTCOMES:
Heart failure quality-of-life | Measured at 1, 6, 12 months
Heart failure-related hospitalizations | Measured at 12 months
Difference between groups for adoption of appropriate self-management knowledge and behaviors | Measured at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mike Pignone, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - University of California - Los Angeles (UCLA), Los Angeles, California
  - University of California at San Francisco, San Francisco General Hospital, San Francisco, California
  - Northwestern Medical Faculty Foundation Clinics & Northwestern Memorial Hospital Chicago, Chicago, Illinois
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- [Background] DeWalt DA, Broucksou KA, Hawk V, Baker DW, Schillinger D, Ruo B, Bibbins-Domingo K, Holmes M, Weinberger M, Macabasco-O'Connell A, Pignone M. Comparison of a one-time educational intervention to a teach-to-goal educational intervention for self-management of heart failure: design of a randomized controlled trial. BMC Health Serv Res. 2009 Jun 11;9:99. doi: 10.1186/1472-6963-9-99. PMID 19519904
- [Background] Baker DW, DeWalt DA, Schillinger D, Hawk V, Ruo B, Bibbins-Domingo K, Weinberger M, Macabasco-O'Connell A, Pignone M. "Teach to goal": theory and design principles of an intervention to improve heart failure self-management skills of patients with low health literacy. J Health Commun. 2011;16 Suppl 3(Suppl 3):73-88. doi: 10.1080/10810730.2011.604379. PMID 21951244
- [Result] Baker DW, Dewalt DA, Schillinger D, Hawk V, Ruo B, Bibbins-Domingo K, Weinberger M, Macabasco-O'Connell A, Grady KL, Holmes GM, Erman B, Broucksou KA, Pignone M. The effect of progressive, reinforcing telephone education and counseling versus brief educational intervention on knowledge, self-care behaviors and heart failure symptoms. J Card Fail. 2011 Oct;17(10):789-96. doi: 10.1016/j.cardfail.2011.06.374. Epub 2011 Jul 23. PMID 21962415
- [Result] Macabasco-O'Connell A, DeWalt DA, Broucksou KA, Hawk V, Baker DW, Schillinger D, Ruo B, Bibbins-Domingo K, Holmes GM, Erman B, Weinberger M, Pignone M. Relationship between literacy, knowledge, self-care behaviors, and heart failure-related quality of life among patients with heart failure. J Gen Intern Med. 2011 Sep;26(9):979-86. doi: 10.1007/s11606-011-1668-y. Epub 2011 Mar 3. PMID 21369770
- [Derived] DeWalt DA, Schillinger D, Ruo B, Bibbins-Domingo K, Baker DW, Holmes GM, Weinberger M, Macabasco-O'Connell A, Broucksou K, Hawk V, Grady KL, Erman B, Sueta CA, Chang PP, Cene CW, Wu JR, Jones CD, Pignone M. Multisite randomized trial of a single-session versus multisession literacy-sensitive self-care intervention for patients with heart failure. Circulation. 2012 Jun 12;125(23):2854-62. doi: 10.1161/CIRCULATIONAHA.111.081745. Epub 2012 May 9. PMID 22572916